CLINICAL TRIAL: NCT03146858
Title: Prolonged Enoxaparin In Primary Percutaneous Coronary Intervention; A Pilot Pharmacodynamic Study
Acronym: PENNY PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STH19752
Record Dates: First submitted 2017-03-27; First posted 2017-05-10 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Primary Percutaneous Coronary Intervention
MeSH Terms: interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: Once patients have been recruited into the trail, they will undertake the first of 4 blood samples. Following the samples the PPCI treatment with begin. The enoxaparin infusion will be set up when the treatment begins. At the end of the PPCI treatment the second blood sample will obtained. The enoxaparin infusion will be commenced after a kidney function check has been performed. The third blood sample will be taken 3 hours into the infusion, and the 4th sample taken at the end of the 6 hour infusion. A 12 hour clinical follow up will then be performed and will mark study completion for the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enoxaparin (Experimental): The patients will receive a 3-6 hour infusion of enoxaparin. The effects of the infusion will be assess when used on patients will acute heart attacks and undergoing emergency treatment with PPCI.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Enoxaparin is an anticlotting treatment that targets the other aspect of clot formation known as the coagulation cascade. Enoxaparin or an alternative is recommended as a single does to support PPCI procedure.

SUMMARY:
Heart attacks are caused by a clot blocking one or more of the heart arteries (coronary arteries). When complete blockage of one of the arteries occurs, emergency treatment to unblock the affected artery and rescue the heart muscle at risk is essential. This is usually achieved by performing an emergency procedure called primary percutaneous coronary intervention (PPCI).

Anticlotting treatment is also necessary to reduce the chances of further heart attacks. As part of standard care, tablets that target small cells called platelets (central to blood clot formation) are given as soon as an acute heart attack is suspected. These tablets include aspirin and ticagrelor/prasufrel. Although both ticgrelor and prasugrel are effective, the onset of action is delayed by up to 8 hours when given in context of an acute heart attack. This delay in onset of action can increase the risk of further heart attacks.

Enoxaparin is an anticlotting treatment that targets the other aspect of clot formation known as coagulation cascade. Enoxaparin or an alternative is recommended as a single does to support the PPCI procedure. The effects of a single shot of enoxaparin do not last long enough to bridge the gap in anticlotting treatment caused by the delayed action of ticagrelor/prasugrel. Since the investigators have realised the delayed onset of action of tablet therapy, the investigators have been using another drug called tirofiban as a drip. Tirofiban blocks platelets effectively, but greatly increases the risk of bleeding events.

The investigators believe that giving enoxaparin as a drip for 3-6 hours (following the single dose) instead of tirofiban, would be sufficient to bridge the gap in anticlotting effect without greatly increasing the risk of bleeding. This is a pilot study to assess the effects of enoxaparin drip in patients presenting with acute heart attacks and undergoing emergency treatment with PPCI.

DETAILED DESCRIPTION:
This is a single centre, pharmacodynamic pilot study of a prolonged enoxaparin infusion following the guideline directed bolus treatment in patients undergoing PPCI conducted at Sheffield Teaching Hospitals NHS Foundation Trust.

Patients admitted to the catheter laboratory or coronary care unit with STEMI and accepted for PPCI will be screened. Those meeting the inclusion criteria will be recruited following angiography. Aspirin is usually administered in the ambulance prior to patient's arrival to hospital and ticagrelor or prasugrel is given as soon as possible on arrival to hospital. This is part of standard clinical care.

The proposed anticoagulant intervention is a parenteral (intra-arterial or intravenous; IA/IV) bolus dose of enoxaparin (0.5 mg/kg) at the time of PPCI followed by an infusion of 0.5 mg/kg over a 6-hour period. In patients with impaired kidney function (eGFR < 30 ml/min), the infusion will be stopped at 3 hours (cumulative dose of 0.75 mg/kg).

Blood samples for anti Xa activity, VerifyNow P2Y12 assay and fibrin clot dynamics will be collected at the following time points:

1. Time point 1 (T1) prior to anticoagulation - at the start of PCI procedure.
2. Time point 2 (T2) at the end of PPCI.
3. Time point 3 (T3) 2-3 hours from the start of enoxaparin infusion.
4. Time point 4 (T4) at the end of enoxaparin infusion. In patients with impaired kidney function (eGFR < 30 ml/min), T3 will be the last blood sample taken (at the end of the infusion).

As PPCI is time critical and delay in treatment can be detrimental to clinical outcome, informed written consent will not be possible prior to the procedure. However, verbal consent using an abbreviated patient information sheet will be obtained prior to enrolment. This will be clearly documented in the patient hospital notes and CRF. As soon as possible after the procedure and whenever possible prior to obtaining T3 blood sample, full written informed consent will be obtained. Blood sampling for T1 and T2 will be done through the arterial sheath and therefore should not cause any significant delay or distress. In the unlikely event where a participant deteriorates and loses capacity during the study, they will be withdrawn from the study but data and blood samples obtained with consent will be retained in the study. In such a case, the treating cardiologist will decide whether to continue with the enoxaparin infusion or not. The consent process will be performed by a qualified medical practitioner according to the principles of Good Clinical Practice (GCP) and the declaration of Helsinki. Following consent, details of patient participation will be sent to their general practitioner.

Clinical outcomes and adverse events will be recorded 12 hours after the end PCI or at the time of transfer to another hospital, whichever comes first. The half-life of enoxaparin is 1-2 hours when given intravenously, and therefore, adverse events are unlikely to arise following the proposed follow-up period.

The primary objective is to assess the pharmacodynamic effect of a prolonged enoxaparin infusion in the context of PPCI. This will be achieved by serial measurements of anti Xa activity.

For inclusion in the study, subjects should fulfil the following criteria:

1. Age ≥ 18
2. Confirmation of the diagnosis of STEMI by the clinical team on the basis of history, ECG changes and angiographic findings
3. Pre-treatment with either ticagrelor or prasugrel
4. Intention to proceed with PPCI
5. Feasibility to obtain informed verbal consent pre PPCI

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Active bleeding that cannot be controlled by local measures
2. Female patients of child bearing age who have not had a sterilisation procedure
3. Patients with end stage renal failure requiring renal replacement therapy
4. Known thrombocytopenia (Platelet count < 100,000/μL)
5. Known history of intracranial haemorrhage
6. Known current treatment with oral anticoagulants
7. Known history of major surgery or trauma or history of GI/GU haemorrhage within the last month
8. Known intracranial malignancy or aneurysm
9. Known allergy to enoxaparin
10. Inability to easily understand verbal information given in English for any reason
11. Inability to give informed consent due to either temporary or permanent mental incapacity

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Confirmation of the diagnosis of STEMI by the clinical team on the basis of history, ECG changes and angiographic findings
* Pre-treatment with either ticagrelor or prasugrel
* Intention to proceed with PPCI
* Feasibility to obtain informed verbal consent pre PPCI

Exclusion Criteria:

* Active bleeding that cannot be controlled by local measures
* Female patients of child bearing age who have not had a sterilisation procedure
* Patients with end stage renal failure requiring renal replacement therapy
* Known thrombocytopenia (Platelet count < 100,000/μL)
* Known history of intracranial haemorrhage
* Known current treatment with oral anticoagulants
* Known history of major surgery or trauma or history of GI/GU haemorrhage within the last month
* Known intracranial malignancy or aneurysm
* Known allergy to enoxaparin
* Inability to easily understand verbal information given in English for any reason
* Inability to give informed consent due to either temporary or permanent mental incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
anti Xa activity change | recruitment, baseline, 3 hrs from baseline, 6 hrs from baseline
  To assess the pharmacodynamic effect of a prolonged enoxaparin infusion in the context.of PPCI. This will be achieved by serial measurements of anti Xa activity.

SECONDARY OUTCOMES:
P2Y12 Inhibition change | recruitment, baseline, 3 hrs from baseline, 6 hrs from baseline
  Assess the level of P2Y12 inhibition in response to oral therapy. This will be achieved by performing the established VerifyNow P2Y12 assay. Although the delay in platelet inhibition is well established now, measuring P2Y12 inhibition is valuable in this case to ensure that adequate inhibition is achieved by the end of enoxaparin infusion. It would also provide useful information in case of complications such as stent thrombosis or bleeding.
Fibrin Clot Formation change | recruitment, baseline, 3 hrs from baseline, 6 hrs from baseline
  Assess the effects of the proposed regimen on fibrin clot formation. This will be done by thromboelastography (TEG) in whole blood and by turbidimetric assay in plasma
Enoxaparin Regimen | within 12 hours from baseline
  Obtain pilot data on the safety of the enoxaparin regimen by assessing bleeding rates 12 hours following PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karunakaran A, Sumaya W, Gunn JP, Morton AC, Storey RF. Contemporary management of ST-segment elevation myocardial infarction. Hosp Pract (1995). 2012 Feb;40(1):224-31. doi: 10.3810/hp.2012.02.963. PMID 22406898
- [Result] Huynh T, Perron S, O'Loughlin J, Joseph L, Labrecque M, Tu JV, Theroux P. Comparison of primary percutaneous coronary intervention and fibrinolytic therapy in ST-segment-elevation myocardial infarction: bayesian hierarchical meta-analyses of randomized controlled trials and observational studies. Circulation. 2009 Jun 23;119(24):3101-9. doi: 10.1161/CIRCULATIONAHA.108.793745. Epub 2009 Jun 8. PMID 19506117
- [Result] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416